CLINICAL TRIAL: NCT05371119
Title: Effects of a Physical Activity Program With Partial Vascular Occlusion on Body Composition, Biomechanics and Walking Energy in Overweight Sedentary Subjects
Brief Title: BFR in Overweight Sedentary Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Gregoire Millet, Professor, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-02081
Record Dates: First submitted 2022-04-19; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Overweight
Keywords: blood flow restriction
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: The procedure will consist of 6 weeks of training with or without partial vascular occlusion (depending on group A or group B) at the rate of 3 sessions per week (for a total of 18 training sessions).
Who Masked: Participant
Masking Description: BFR inflated 20 mmHg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (Experimental): Use of the BFR cuff during the training intervention
  Interventions: Other: Exercise Intervention
- control (Active Comparator): No use of inflated cuff
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Training with light load with blood flow restriction (BFR)

SUMMARY:
This project should allow the investigators to observe the effects of low load training under partial vascular occlusion (BFR) in comparison with resistance training at low load without partial vascular occlusion in sedentary people overweight on parameters : decrease in fat mass; increase in muscle mass 79; muscle strength; decrease in the energy cost of walking; increase in preferred walking speed; improvement in walking pattern in patients overweight. Training under partial vascular occlusion should facilitate physical activity in overweight people as it can be just as effective as a "classic" type training with heavy loads. Thus, this device could allow people for who wear heavy loads can present an obstacle to physical activity to feel more involved in the physical activity programs offered in medical or sports centers.

DETAILED DESCRIPTION:
The main objective of this study is to observe the effects of low load training under vascular occlusion (BFR) compared with low load resistance training without vascular occlusion in overweight sedentary people on parameters such as: decrease in fat mass; lower blood sugar levels as well as lower blood triglycerides and cholesterol levels; increased muscle mass; muscle strength; the reduction of the energy cost of walking; increasing the preferred walking speed; improving the walking pattern in overweight patients.

3.2 Primary and secondary endpoints

The first hypothesis is that the BFR drive will be effective in improving walking economy (thus reducing the energy cost of walking) and increasing the preferred walking speed, by improving walking patterns.

The second hypothesis is that BFR training makes it possible to modify the body composition in a slight way and to promote the gain of muscle strength in overweight individuals who do not practice physical activity beforehand. In addition, blood tests will show a decrease in blood sugar, blood triglyceride levels and cholesterol.

3.3 Study design

This single-center project aims to test the effects of low-load training under partial vascular occlusion (BFR) compared to low-load resistance training without vascular occlusion in overweight sedentary people. The main expected effects are a decrease in fat mass, an increase in muscle mass and strength, a decrease in the energy cost of walking as well as an increase in preferential walking speed. This project is part of a continuity of research in a public health context in order to propose adapted and effective physical activity programs for an overweight population unable to train with heavy loads.

ELIGIBILITY:
Inclusion Criteria:

* IMC between 25 and 35
* vaccin against Covid-19

Exclusion Criteria:

hypertension diabete

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
DEXA technology | One week before intervention
  Body composition assessment: relative lean and fat mass in all body segments
DEXA technology | One week following the training intervention
  Body composition assessment: relative lean and fat mass in all body segments
Evaluation of muscle strength from an isokinetic device | One week before intervention
  eccentric and concentric peak torque of the knee extensor muscles
Evaluation of muscle strength from an isokinetic device | One week following the training intervention
  eccentric and concentric peak torque of the knee extensor muscles
Evaluation of the preferential speed of walking in an ecological situation | One week before interventionn
  using of a treadmill with measurement of the ground reaction forces
Evaluation of the preferential speed of walking in an ecological situation | One week following the training intervention
  using of a treadmill with measurement of the ground reaction forces
Analysis of the biomechanics of walking on a treadmill instrumented with power platforms. | One week before intervention
  calculation of the mechanical work
Analysis of the biomechanics of walking on a treadmill instrumented with power platforms. | One week following the training intervention
  calculation of the mechanical work
Evaluation of the energy cost of walking | One week before intervention
  on a treadmill, by indirect calorimetry with gaz exchanges
Evaluation of the energy cost of walking | One week following the training intervention
  on a treadmill, by indirect calorimetry with gaz exchanges

CONTACTS AND LOCATIONS:
Locations (1):
- ISSUL, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No